CLINICAL TRIAL: NCT07095738
Title: Textural Analysis and Effect of ROI Size on Infrared Thermography in Athletes With Patellar Tendinopathy. A Cross-sectional Study
Brief Title: Textural Analysis and Effect of ROI Size on Infrared Thermography in Athletes With Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Clinical Professor, Cardenal Herrera University
Other Study IDs: CE111803
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Patellar Tendinopathy; Diagnostic Accuracy; Infrared Thermography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- athletes with unilateral PT: diagnosed through a combination of clinical criteria, specific functional tests, and ultrasound evaluation. Additional inclusion criteria for this group include a symptom evolution time of more than 3 months, a VISA-P score of less than 80, and the performance of a differential diagnosis to rule out other potential causes of anterior knee pain
  Interventions: Diagnostic Test: thermal images (IT)
- healthy volunteer athletes: recruited under the inclusion criteria of no previous history of PT and a VISA-P score of 100
  Interventions: Diagnostic Test: thermal images (IT)

INTERVENTIONS:
Diagnostic Test: thermal images (IT) — The IT images were recorded with an OPTRIS PI 450 IRT camera coupled to Optris PI Connect Software (Germany). The IRT camera has a Noise Equivalent Temperature Difference <40 mK with 38º x 29º FOV, a wide range of temperature from -20°C to +100°C, spectrum range of 7.5-13 μm, focal plane array sensor size of 382 × 288 pixels, emissivity set at 0.98 and a measurement uncertainty of ± 2% of the overall temperature reading. The size of the capture frame will be 55.4 × 40.63 cm (1.5 mm/px).

SUMMARY:
Patellar tendinopathy (PT) is a common knee disorder, particularly among elite athletes, with a reported prevalence of approximately 14.2%. Athletes affected by PT may experience persistent pain, functional impairment, reduced quality of life, decreased physical performance, and even premature career termination. Diagnosing PT remains challenging due to the absence of a gold standard diagnostic method. Although imaging techniques such as ultrasonography (US) and magnetic resonance imaging (MRI) can aid in confirming the diagnosis and assessing severity, MRI is costly and less accessible, and US shows poor correlation with clinical symptoms. Consequently, diagnosis largely relies on clinical examination and medical history. Infrared thermography (IT) has emerged as a potential alternative imaging technique, offering a low-cost, reliable, and non-invasive method to detect thermal asymmetries indicative of underlying pathologies. Technological advancements have enhanced the precision of IT, reducing the thermal asymmetry threshold from 2-3 ºC in the 1970s to 0.5 ºC in current knee assessments. First-order statistics, such as mean gray intensity, and second-order features based on the gray-level co-occurrence matrix (GLCM), have been extensively used in medical image analysis, including IT, to quantify structural and textural characteristics. The size of the region of interest (ROI) is also a critical factor in thermal and texture analyses, as it can influence sensitivity and diagnostic accuracy. Given these considerations, the objectives of this study were: (1) to evaluate differences in thermal and GLCM-based textural features between athletes with PT and healthy controls; (2) to compare the diagnostic performance of IT and GLCM features applied to thermographic images; and (3) to identify the most appropriate ROI size for optimal characterization of PT using both thermal and textural analysis.

ELIGIBILITY:
Inclusion Criteria:

* Specific functional tests.
* Ultrasound evaluation.
* Symptom evolution time of more than 3 months.
* A VISA-P score of less than 80.
* The performance of a differential diagnosis to rule out other potential causes of anterior knee pain.

Exclusion Criteria:

* Lower limb pathology.
* Nerve or vascular disorder, or skin lesion in the knee area that could alter thermal information in the patellar tendon region.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be instructed not to engage in physical exercise; not to drink alcohol, coffee, or energy drinks 12 hours prior to measurements; not to smoke in the 6 hours prior to measurements; not to apply creams or lotions to their legs to avoid altering skin emissivity; to report any medication or treatments they were taking; and to try to avoid altering their rest and meal habits. These requirements minimise the influence of individual extrinsic factors on the IT results.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Textural analysis based on the Gray-Level Co-occurrence Matrix (GLCM) | baseline
  GLCM relies on the angular relationship between neighboring pixels and the distance between them. relies on the angular relationship between neighboring pixels and the distance between them.
Energy or angular second moment (ASM) | baseline
  ASM Measures the uniformity or regularity in the distribution of image values. Higher values indicate greater uniformity in the image.
Homogeneity or inverse difference moment (IDM) | baseline
  IDM reflects the homogeneity of image composition, associated with pixel pairs. Homogeneous images with minimal variations produce high IDM values
Contrast (CON) | baseline
  CON represents the degree of local variations in gray levels within the image.If the variation increases, the contrast increases.
Textural correlation (TCOR) | baseline
  TCOR expresses linear dependencies between gray levels in the image. Regions with similar gray levels tend to exhibit higher values.
Entropy (ENT) | baseline
  Indicates the level of disorder within the image. Homogeneous images result in lower entropy values

SECONDARY OUTCOMES:
Age (years) | baseline
Sex | baseline
Body Mass index (BMI) | baseline
  kg/m²
time of evolution (months) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ceu Cardenal Herrera University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data associated with this paper will be available in the Zenodo repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: baseline

REFERENCES:
- See also: Group investigation — https://www.uchceu.es/grupos-lineas-investigacion/fisioterapia-activa-terapia-manual-y-analisis-de-imagen-fami

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT07095738/Prot_SAP_ICF_000.pdf